CLINICAL TRIAL: NCT02455232
Title: Determine the Main Muscle Participant in the Deformation of the Elbow in Hemiplegic Patients
Acronym: FLEXELBOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-A00444-45
Record Dates: First submitted 2015-05-07; First posted 2015-05-27 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Hemiplegia
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hemiplegic patient (Experimental): muscle participation in upper limb spasticity
  Interventions: Procedure: upper limb muscle block; Drug: 4cc of lidocaïne®

INTERVENTIONS:
Procedure: upper limb muscle block
Drug: 4cc of lidocaïne®

SUMMARY:
The aim of this study is to determinate what are the main muscles regularly involved in the spastic pattern in flexion of the elbow using the selective motor nerve blocks of the elbow flexors. Three selective motor block nerves will be carry out in order to assess the gain of the range of motion (passive and active) of the elbow after each Motor Block Nerve.

DETAILED DESCRIPTION:
To assess the impact of selective motor block nerves (successively brachialis motor branch, radialis motor nerve and musculocutaneous motor branch) on passive and active ranges of motion of the elbow in stroke patients with spastic flexion pattern.

Procedure: Following the morphological landmarks already described, the brachialis motor nerve of 30 patients was blocked with 4cc of lidocaïne® 1% (electro stimulation 0.8 to 1mA) (ref). Twenty minutes after the injection, the measurement of the degree of the spasticity, the passive angle in extension and the active range of motion in flexion of the elbow were performed. Then the radialis motor nerve block was performed (at the union of the median third and lower third of the arm, medial view, 3 finger widths above the medial epicondyle) using the same procedure, in order to block the brachioradialis and the brachialis in case of double innervation. Twenty minutes after the injection, the measurement of the passive and active ranges of motion of the elbow was performed. At the end the musculocutaneous motor block nerve was performed (proximal quarter of the arm, medial view, at the base of the inferior limit of the pectoralis major and along the biceps brachii tendon) in order to make the final difference with muscle contracture if it existed a doubt.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* Hemiplegic patient with spasticity and deformation of elbow

Exclusion Criteria:

* pregnant woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
angles of elbow as measured by means of a goniometer | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: François Genet, PhD, Principal Investigator — Centre d'Investigation Clinique et Technologique 805
Locations (1):
- Hopital Raymond Poincaré, Garches, Garches, France